

NCT Number: NCT06493214

Document Date: 6/27/2024

## Assent to Participate in a Research Study (8-12 year olds)

We want to tell you about a research study we are doing and see if you want to take part in it. Research is a way to learn more about something. If you have any questions about what we are telling you, just ask us! You can ask us questions now and anytime you think of them.

We want to find out what resources will help kids, just like you, do a physical activity program at home. We will be trying a few different resources designed for you, your parent (or guardian), and your family.

You are being asked to be in this research study because you are a child that is 8-12 years old. For you to join, both you and your parent (or guardian) must agree to you being in it. It is the adult's job to make sure this study is okay for you. But it is still up to you if you *want* to do it. Parents and children say "no" for different reasons. If you say "no," that's okay, and you won't be treated differently. You can also change your mind at any point!

If you decide to join this study and your parent (or guardian) says "yes", here is what you will do:

- We will ask you to do 3, 8-minute physical activity videos in your home, 5-days per week for 60 days (3 months). The videos have exercises like jumping jacks and running in place and others like push-ups and squats. Your goal is to do all 3 videos each day, but it's okay if you are unable to do that each day. These videos are online and so you can do them at home!
- You will be asked to write down how many videos you do each day and how hard you felt like you were working during them.
- We will ask you to wear a physical activity watch (Fitbit) around your wrist to keep track of how much you move during the physical activity videos.
- You may also receive resources to help you do these physical activity videos.
- We will ask you to answer some questions about your health, emotions, enjoyment of physical activity, and daily physical activity at the beginning and end of the study.

We do not know for sure if you will be helped by being in this study, but we might learn what will help other children with doing physical activity at home. Some of the benefits you could gain are:

- You will get to do fun physical activity videos at home!
- You will gain access to virtual physical activity videos you can do, even after the study ends.

Some of the things you may feel during this study are:

- You might not like every video you do (and that's okay! Be sure to let us know which ones you like and don't like).
- You may feel tired or have sore msucles from exercising. Overtime, you
  may become more fit and be able to bounce back from being tired quicker.
- You may feel annoyed with wearing the Fitbit watch.
- You may feel uncomfortable with some of the questions we ask. You can can skip any questions that you do not want to answer, whatever the reason, and you do not have to tell us why.

Your information will be kept secret and safe, and your name will not be on your results. Only the research team will know your results and have access to your data.

You should also know that we have to report certain types of information. If you tell us, or we learn something that makes us believe that you or others have been, or may be, physically harmed, we may be required to report that information to the right people.

If you complete the full study, you will receive a new Fitbit valued up to \$75, a jump rope and a water bottle. If you complete two months of the study, you will receive a jump rope and a water bottle. If you complete one month of the study, you will receive a jump rope.

| researcher to explain | or someone has read it to me. If I did not understand something, I asked the it to me. I can always ask the researcher a question about the study if I don't ing. I will be given a copy of this form. |
|---|---|
| Please check one be | ox: |
| ☐ YES, I wa | ant to be in this study and I know I can change my mind later. |
| | not want to be in this study. |
| Child's Name (print legal name): | |
| Child's Signature: | |
| Date of signature: | Age # |

The following should be completed by the study member conducting the assent process if the child agrees to be in the study. Check all that apply.

- € The child is capable of reading and understanding the assent form and has signed above as documentation of assent to take part in this study.
- € The child is not capable of reading the assent form, but the information was verbally explained to him/her. The child signed above as documentation of assent to take part in this study.
- € The child had ample opportunity to have his or her questions answered.

| Printed name of person obtaining agreement: |
|---------------------------------------------|
| Signature of person obtaining agreement: |
| Date of signature: |